CLINICAL TRIAL: NCT04478487
Title: TITLE OF STUDY: Safety and Efficacy of a Novel Human Milk-based Human Milk Fortifier in Very Low Birth Weight Infants
Brief Title: Novel Human Milk Based Human Milk Fortifier
Acronym: MHMHMF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwest Health (Other)
Collaborators: Neolac Inc dba Medolac Laboratories (Industry)
Responsible Party: Principal Investigator, Sameer Wagle, MD, Medical Director, NICU, Northwest Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC-2018-01
Record Dates: First submitted 2020-06-18; First posted 2020-07-20 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Intervention Model Description: This is a non-controlled observational trial using objective measures (body weight) to assess the support of growth and tolerance of a new fortifier based on human milk, thereby enabling an exclusive human milk diet for VLBW infants in the NICU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental): all preterm infants ≤ 32 weeks and 0 days gestational age (GA) with a birth weight 700 g to 1500 g at the hospital, who are enterally fed human milk in the neonatal intensive care unit (NICU) for at least 7 days. Various blending ratios of the fortifier with either the mother's expressed milk or donor milk will be used to deliver macro and micronutrients based on established guidelines to be adjusted according to the infant's tolerance for volume and calories. The estimated time for each subject's participation is approximately from 1 week through 8 weeks, depending on the weight and age at enrollment. Historic control cases treated by another human milk based human milk fortifier will be obtained from medical records, matched on birth weight and gender, with sample size twice (n=80) that of the study population.
  Interventions: Dietary Supplement: Medolac human milk based human milk fortifier (MHMHMF)

INTERVENTIONS:
Dietary Supplement: Medolac human milk based human milk fortifier (MHMHMF) — MHMHMF is admixed with expressed or donor human milk in graded doses according to tolerated feed volume according to established guidelines and maintain adequate micronutrient levels.
  Other Names: exclusive human milk diet for VLBW infants

SUMMARY:
The primary objective is to assess weight gain of VLBW infants fed human milk supplemented with a novel human milk-based fortifier, in comparison to use of other fortifiers (historic controls).

DETAILED DESCRIPTION:
Background Once feeding low birthweight (LBW) or very low birthweight (VLBW) infants was primarily by commercial specialty formulas. As public health emphasis on breastfeeding increased awareness and prevalence of breastfeeding, the use of human milk in the Neonatal Intensive Care unit (NICU) became more common. However, despite the fact that milk from mothers delivering prematurely has higher nutritional content than milk from mothers delivering at term, mainly in protein and fat, thus calories, nutrient intake from human milk alone is not sufficient to satisfy the nutrition of the LBW or VLBW infants and support intrauterine growth rates. Low birth weight infants have faster growth when fed preterm formula compared to when they are breastfed. Consequently, human milk fortifiers (HMF) with an emphasis on protein and caloric density (to accommodate small gastric volume among these babies) but with major minerals and selected micronutrients were developed as supplements to admix with human milk for feeding preterm infants. HM fortifiers were initially based on cows milk proteins and were manufactured as either powders or liquids, the latter having the benefit of being sterile, avoiding the risk of contamination by bacterial contaminants in powders, eg, cronobacter sakazakii. Attention to early life nutrition has reduced the prevalence of growth restricted infants at discharge.

Protein Increased protein in fortifiers in LBW feeds directly improves weight gain, and early introduction of fortifiers may mitigate typical protein intake shortfall that is seen during the transition from parenteral to enteral feeding. The highest useful protein level may have been determined.Growth of VLBW infants fed primarily breast milk supplemented with bovine milk fortifier to obtain 4.3 g protein/kg/d was not improved over infants whose milk fortification was 3.7 g/kg/d; both groups nearly achieved intrauterine growth rates. Breast milk comprised 92 and 94% of total food intake and average daily weight gains were 16.3 g/kg and 16.0 g/kg in the lower and higher protein groups, respectively. Length and head circumference gains were similar between groups. In one study bovine based fortifier providing total protein at a yet higher level of 4.6- 5.4 g/kg/d reported improved length gain, but not weight gain.

Other variations of protein presentation also have been reported. Liquid HMF made with extensively hydrolyzed protein at 3.6g/100 kcal gave slightly better weight gain than powdered intact protein containing 3 g protein/100 kcal. A new powdered presentation using partially hydrolysed whey protein at 16% higher total protein content than the commercial product with intact protein gave improved weight gain. In addition to the protein content, processing is important. Acidified liquid fortifier-fed infants fared poorer than infants fed neutral pH sterilized HMF even though the acidified formula had higher protein intake (4.2 g/kg) than the sterilized (3.7 g/kg).

None of these studies assessed the effects of different levels of human milk protein, but they suggest attention be paid to achieving protein targets; that liquids may be preferred over powders, and that sterilized neutral pH products are preferable to acidified products.

Necrotizing enterocolitis (NEC) One study created awareness about the value of feeding exclusive human milk in the NICU and reported that there was no difference in growth between VLBW infants fed mothers own milk supplemented with a fortifier derived from donor human milk or when a fortifier based on bovine milk was used, though the exclusively human milk diet resulted in fewer cases of NEC and NEC requiring surgical intervention. Subsequently, another study reported feeding with a fortifier based on human milk reduced days of parenteral nutrition (p=0.04), trend toward all NEC (p= 0.08) and reduced surgical NEC (p=0.04) when compared to fortification with preterm bovine milk based formula. Others report the timing of onset of NEC was delayed and incidence of late onset NEC (after 7 feeding days) and incidence of sepsis was significantly reduced among infants fed exclusive human milk diets compared to an earlier cohort of infants supplemented with bovine products; however, respiratory distress syndrome and use of surfactants was more common among the exclusive human milk cohort, and infants fed bovine products were more commonly discharged to home. A 2014 Cochrane review of 9 studies found an increased risk of NEC among infants fed preterm formulas. This conclusion has been supported by recent retrospective studies, and extending benefit of exclusive human milk diets to reduced risk of bronchopulmonary dysplasia (BPD) and retinopathy of prematurity (ROP) in addition to NEC .

The value of exclusive human milk feeding also has been explored regarding growth. Questions of the relative value of mother's own milk compared to donor human milk, the form of fortifier (powder v liquid, v acidified liquid), the level of protein, and the source of protein (bovine or human) have been explored. A study reported that infants fed >75% donor milk had higher risk of small for gestational age (SGA) compared to those fed their own mothers milk. Donor milk fed infants had lower weight gain than infants fed either moms own milk or preterm formula possibly because of lower nutrient content of donor milk. In contrast, VLBW infants fed their own mother's milk fortified alternatively with donor milk or preterm formula grew better (weight gain from birth to discharge) as the proportion of diet as breast milk increased from <25%, 25-50%, to > 75% of total intake. A retrospective analysis among extremely low birthweight infants (ELBW) exclusively human milk diets reported a comparable growth and neurodevelopment as infants fed bovine milk based fortifiers.

Consequently, there is good evidence that fortification of human milk is needed to support growth of LBW and VLBW infants, that higher protein up to about 4.3 g/kg/d supports more rapid growth, and that risk of NEC and other diseases affecting LBW infants is less when LBW infants are fed exclusive human milk diets. The difficulties have been to obtain liquid fortifier derived from human milk, and evaluate its use at the protein concentrations that have been evaluated using bovine-based products. This study addresses these two needs: a sterile liquid fortifier derived from human milk is evaluated at protein intakes recommended by the European Society for Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN), 4.0-4.5 g/kg/d for infants less than 1000g, and 3.5-4.0 g/kg for infants 1000-1800g.

Summary of Nonclinical Experience with MHMHMF The preclinical experience with this particular fortifier is limited to analytical evaluation. There are no suitable animal models sensitive to testing the biological source of the protein, and no alternative method for assessing growth of infants fed a human protein-based fortifier than clinical study. The protein quality of the processed protein has been established by amino acid analysis to be close to the native protein, with up to a 15% decrease in available lysine, probably due to Maillard reaction with lactose. The fortifier, even at its lowest recommended use rate represents more than a 2-fold increase in all amino acids when compared to raw breast milk, we are not concerned about protein quality with our manufacturing process. Additionally, the composition of the blended fortifier exceeds Codex reference for protein quality for infant formula and formulas for special medical purposes intended for infants.

Summary of Clinical Experience Medolac has processed donor whole human milk for feeding LBW infants for some years. More recently Medolac has applied standard dairy processes to partition milk into milk fat and skim fractions, and to enrich the protein content. The processes have allowed the development of high protein human milk fortifier. Supplementation of the high protein fraction with vitamins and minerals has resulted in a novel human milk based human milk fortifier for fortification of human milk-fed VLBW infants. This is the first clinical evaluation of the MHMHMF fortifier. Only one other fortifier derived from human milk is available commercially (Prolacta). Reports on its use have been published showing reduced days of parenteral nutrition (p=0.04), trend toward all NEC (p= 0.08) and reduced surgical NEC (p=0.04) and rescue from failure after use of bovine based fortifiers.

Description of Investigational Product The investigational product is manufactured from whole human breast milk with the addition of selected vitamins and minerals. The source of human milk is full lactation, full term donor milk from Mothers Milk Cooperative (Boulder City, NV), collected according to stringent blood screening criteria and quality control procedures, including microbiological evaluation, nutritional composition and chemical analyses. A fractionated, concentrated product is created by first delipidating then filtering through ultrafiltration (UF) membranes to selectively concentrate protein with loss of low molecular weight components such as lactose and minerals. Fat, selected minerals, and vitamins are added to the protein enriched fluid to reach a standard ratio. It is then packaged and processed by heat to achieve commercial sterility, granting room temperature storage with extensive shelf-life.

Various blending ratios of the fortifier with either the mother's expressed milk or donor milk can be used to deliver varying concentrations of vitamins, minerals, and macronutrients enabling nutrient delivery to be adjusted according to the infant's tolerance for volume and calories.

Blending ratios are illustrated in the table below. Simple blending of 50:50 results in a high protein, fat enriched fortifier having a caloric density of 27 kcal/ounce with protein provided at 3.0g/100 milliliters (mL). When this fortifier is mixed in a 1:2 ratio, the resulting caloric density is 25 kcal/oz and protein is provided at 2.4 g/100 ml; when this fortifier is mixed in a 1:3 ratio, the resulting caloric density is 23.6 kcal/oz and protein is provided at 2.07 g/100 ml; Similarly, other nutrients are delivered as a function of the ratio of MHMHMF to human milk.

The primary objective for growth with this fortifier is the delivery of protein and calories, however we recognize that some vitamins are cofactors of enzymes involved in protein and energy metabolism. Some minerals such as zinc is variable in human milk, so was selected for addition. Other vitamins and minerals such as iron are generally monitored while others such as copper, vitamin A, and niacin are not considered limiting in human milk. In addition, heat processing used to achieve commercial sterility degrades some vitamins, making separate administration desirable. For these reasons the MHMHMF is not comprehensive in its delivery of vitamins and minerals which have been shown to be essential for nutrition. Infants should be monitored for adequate nutrition and additional fortification given as needed.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight between 750 g-1500 g.
* ≤ 32 weeks gestational age at birth. GA will be determined by an ultrasound scan or the neonatologist's estimate, with consideration to maternal date.
* Subject has been classified as appropriate for GA (AGA).
* Enteral feeding of human milk must be initiated by 21 days of life for infants with a birthweight of 750-1000 g (birth date is day of life 0) and initiated by 14 days of life for infants with a birthweight of 1.0 - 1.5 kg birthweight.
* Mother agrees to feed the infant human milk as the exclusive feeding during the study period. Human milk may be mothers own or donor milk, plus MHMHMF.
* Singleton or twin births only.

Exclusion Criteria:

* Serious congenital abnormalities or underlying disease that may affect growth and development.
* 5 minute APGAR: 5 4.
* Steroids used within the past 5 days
* Grade Ill or IV periventricular/ intraventricular hemorrhage (PVH/IVH).
* Maternal cocaine, alcohol or opioid abuse during pregnancy or currently or if the mother or infant is currently receiving treatment for HIV infection.
* Infant major surgery (intra-thoracic or intra-abdominal procedures or other surgery requiring general anesthesia).
* Asphyxia defined as progressive hypoxemia and hypercapnia with significant metabolic acidemia characterized by APGAR score <3 at 10 minutes, seizures within the first 12 hours of life, or a cord blood gas < 7.0 and seizures and/or severe tonic abnormalities in the first 12 hours of life.
* Infant has any other condition that, in the opinion of the investigator, compromises the ability to draw inference about the ability of the MHMHMF to support growth.

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
weight gain (gm/kg/day) | Daily from first day of enrollment until 36 weeks post menstrual age or discharge
  Weights.

SECONDARY OUTCOMES:
length increment (cm/kg/day) | Weekly until 36 weeks post menstrual age or discharge
  length
Head Circumference increment (cm/kg/day) | Weekly until 36 weeks post menstrual age or discharge
  Head circumference
Volume of Fortifier | Daily until 36 weeks post menstrual age or discharge
  Total intake of formula and fortifier
Morbidity | weekly until 36 weeks post menstrual age or discharge
  Adverse Events-necrotizing enterocolitis, retinopathy of prematurity and bronchopulmonary dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Fels, Study Director — Medolac Laboratories
Locations (1):
- Willow Creek Women's Hospital, Johnson, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agostoni C, Buonocore G, Carnielli VP, De Curtis M, Darmaun D, Decsi T, Domellof M, Embleton ND, Fusch C, Genzel-Boroviczeny O, Goulet O, Kalhan SC, Kolacek S, Koletzko B, Lapillonne A, Mihatsch W, Moreno L, Neu J, Poindexter B, Puntis J, Putet G, Rigo J, Riskin A, Salle B, Sauer P, Shamir R, Szajewska H, Thureen P, Turck D, van Goudoever JB, Ziegler EE; ESPGHAN Committee on Nutrition. Enteral nutrient supply for preterm infants: commentary from the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):85-91. doi: 10.1097/MPG.0b013e3181adaee0. PMID 19881390
- [Background] Cacho NT, Parker LA, Neu J. Necrotizing Enterocolitis and Human Milk Feeding: A Systematic Review. Clin Perinatol. 2017 Mar;44(1):49-67. doi: 10.1016/j.clp.2016.11.009. Epub 2016 Dec 24. PMID 28159209
- [Background] Chowning R, Radmacher P, Lewis S, Serke L, Pettit N, Adamkin DH. A retrospective analysis of the effect of human milk on prevention of necrotizing enterocolitis and postnatal growth. J Perinatol. 2016 Mar;36(3):221-4. doi: 10.1038/jp.2015.179. Epub 2015 Dec 3. PMID 26633147
- [Background] Colacci M, Murthy K, DeRegnier RO, Khan JY, Robinson DT. Growth and Development in Extremely Low Birth Weight Infants After the Introduction of Exclusive Human Milk Feedings. Am J Perinatol. 2017 Jan;34(2):130-137. doi: 10.1055/s-0036-1584520. Epub 2016 Jun 20. PMID 27322667
- [Background] Colaizy TT, Carlson S, Saftlas AF, Morriss FH Jr. Growth in VLBW infants fed predominantly fortified maternal and donor human milk diets: a retrospective cohort study. BMC Pediatr. 2012 Aug 17;12:124. doi: 10.1186/1471-2431-12-124. PMID 22900590
- [Background] Cristofalo EA, Schanler RJ, Blanco CL, Sullivan S, Trawoeger R, Kiechl-Kohlendorfer U, Dudell G, Rechtman DJ, Lee ML, Lucas A, Abrams S. Randomized trial of exclusive human milk versus preterm formula diets in extremely premature infants. J Pediatr. 2013 Dec;163(6):1592-1595.e1. doi: 10.1016/j.jpeds.2013.07.011. Epub 2013 Aug 20. PMID 23968744
- [Background] Fenton TR, Kim JH. A systematic review and meta-analysis to revise the Fenton growth chart for preterm infants. BMC Pediatr. 2013 Apr 20;13:59. doi: 10.1186/1471-2431-13-59. PMID 23601190
- [Background] Gidrewicz DA, Fenton TR. A systematic review and meta-analysis of the nutrient content of preterm and term breast milk. BMC Pediatr. 2014 Aug 30;14:216. doi: 10.1186/1471-2431-14-216. PMID 25174435
- [Background] Hair AB, Peluso AM, Hawthorne KM, Perez J, Smith DP, Khan JY, O'Donnell A, Powers RJ, Lee ML, Abrams SA. Beyond Necrotizing Enterocolitis Prevention: Improving Outcomes with an Exclusive Human Milk-Based Diet. Breastfeed Med. 2016 Mar;11(2):70-4. doi: 10.1089/bfm.2015.0134. Epub 2016 Jan 20. PMID 26789484
- [Background] Hay WW, Ziegler EE. Growth failure among preterm infants due to insufficient protein is not innocuous and must be prevented. J Perinatol. 2016 Jul;36(7):500-2. doi: 10.1038/jp.2016.85. No abstract available. PMID 27339826
- [Background] Herrmann K, Carroll K. An exclusively human milk diet reduces necrotizing enterocolitis. Breastfeed Med. 2014 May;9(4):184-90. doi: 10.1089/bfm.2013.0121. Epub 2014 Mar 3. PMID 24588561
- [Background] Horbar JD, Ehrenkranz RA, Badger GJ, Edwards EM, Morrow KA, Soll RF, Buzas JS, Bertino E, Gagliardi L, Bellu R. Weight Growth Velocity and Postnatal Growth Failure in Infants 501 to 1500 Grams: 2000-2013. Pediatrics. 2015 Jul;136(1):e84-92. doi: 10.1542/peds.2015-0129. PMID 26101360
- [Background] Kim JH, Chan G, Schanler R, Groh-Wargo S, Bloom B, Dimmit R, Williams L, Baggs G, Barrett-Reis B. Growth and Tolerance of Preterm Infants Fed a New Extensively Hydrolyzed Liquid Human Milk Fortifier. J Pediatr Gastroenterol Nutr. 2015 Dec;61(6):665-71. doi: 10.1097/MPG.0000000000001010. PMID 26488118
- [Background] Kim EJ, Lee NM, Chung SH. A retrospective study on the effects of exclusive donor human milk feeding in a short period after birth on morbidity and growth of preterm infants during hospitalization. Medicine (Baltimore). 2017 Sep;96(35):e7970. doi: 10.1097/MD.0000000000007970. PMID 28858132
- [Background] Kumar N, Monga R, Sampath V, Ehrhart B. Prospective Comparison of Enfamil and Similac Liquid Human Milk Fortifier on Clinical Outcomes in Premature Infants. Am J Perinatol. 2017 Dec;34(14):1411-1416. doi: 10.1055/s-0037-1603940. Epub 2017 Jun 21. No abstract available. PMID 28637062
- [Background] Liu TT, Dang D, Lv XM, Wang TF, Du JF, Wu H. Human milk fortifier with high versus standard protein content for promoting growth of preterm infants: A meta-analysis. J Int Med Res. 2015 Jun;43(3):279-89. doi: 10.1177/0300060515579115. Epub 2015 May 8. PMID 25956156
- [Background] Maas C, Mathes M, Bleeker C, Vek J, Bernhard W, Wiechers C, Peter A, Poets CF, Franz AR. Effect of Increased Enteral Protein Intake on Growth in Human Milk-Fed Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2017 Jan 1;171(1):16-22. doi: 10.1001/jamapediatrics.2016.2681. PMID 27893064
- [Background] Madore LS, Bora S, Erdei C, Jumani T, Dengos AR, Sen S. Effects of Donor Breastmilk Feeding on Growth and Early Neurodevelopmental Outcomes in Preterm Infants: An Observational Study. Clin Ther. 2017 Jun;39(6):1210-1220. doi: 10.1016/j.clinthera.2017.05.341. Epub 2017 May 30. PMID 28576299
- [Background] McGuire W, Anthony MY. Formula milk versus preterm human milk for feeding preterm or low birth weight infants. Cochrane Database Syst Rev. 2001;(3):CD002972. doi: 10.1002/14651858.CD002972. PMID 11687034
- [Background] Olsen IE, Harris CL, Lawson ML, Berseth CL. Higher protein intake improves length, not weight, z scores in preterm infants. J Pediatr Gastroenterol Nutr. 2014 Apr;58(4):409-16. doi: 10.1097/MPG.0000000000000237. PMID 24231639
- [Background] Rigo J, Hascoet JM, Billeaud C, Picaud JC, Mosca F, Rubio A, Saliba E, Radke M, Simeoni U, Guillois B, de Halleux V, Jaeger J, Ameye L, Hays NP, Spalinger J. Growth and Nutritional Biomarkers of Preterm Infants Fed a New Powdered Human Milk Fortifier: A Randomized Trial. J Pediatr Gastroenterol Nutr. 2017 Oct;65(4):e83-e93. doi: 10.1097/MPG.0000000000001686. PMID 28727654
- [Background] Sandhu A, Fast S, Bonnar K, Baier RJ, Narvey M. Human-Based Human Milk Fortifier as Rescue Therapy in Very Low Birth Weight Infants Demonstrating Intolerance to Bovine-Based Human Milk Fortifier. Breastfeed Med. 2017 Nov;12(9):570-573. doi: 10.1089/bfm.2017.0017. Epub 2017 Aug 4. PMID 28777664
- [Background] Shah SD, Dereddy N, Jones TL, Dhanireddy R, Talati AJ. Early versus Delayed Human Milk Fortification in Very Low Birth Weight Infants-A Randomized Controlled Trial. J Pediatr. 2016 Jul;174:126-131.e1. doi: 10.1016/j.jpeds.2016.03.056. Epub 2016 Apr 23. PMID 27112041
- [Background] Sisk PM, Lovelady CA, Dillard RG, Gruber KJ, O'Shea TM. Early human milk feeding is associated with a lower risk of necrotizing enterocolitis in very low birth weight infants. J Perinatol. 2007 Jul;27(7):428-33. doi: 10.1038/sj.jp.7211758. Epub 2007 Apr 19. PMID 17443195
- [Background] Spiegler J, Preuss M, Gebauer C, Bendiks M, Herting E, Gopel W; German Neonatal Network (GNN); German Neonatal Network GNN. Does Breastmilk Influence the Development of Bronchopulmonary Dysplasia? J Pediatr. 2016 Feb;169:76-80.e4. doi: 10.1016/j.jpeds.2015.10.080. Epub 2015 Nov 25. PMID 26621048
- [Background] Sullivan S, Schanler RJ, Kim JH, Patel AL, Trawoger R, Kiechl-Kohlendorfer U, Chan GM, Blanco CL, Abrams S, Cotten CM, Laroia N, Ehrenkranz RA, Dudell G, Cristofalo EA, Meier P, Lee ML, Rechtman DJ, Lucas A. An exclusively human milk-based diet is associated with a lower rate of necrotizing enterocolitis than a diet of human milk and bovine milk-based products. J Pediatr. 2010 Apr;156(4):562-7.e1. doi: 10.1016/j.jpeds.2009.10.040. Epub 2009 Dec 29. PMID 20036378
- [Background] Taylor C. Health Professionals Letter on Enterobacter sakazakii Infections Associated With the Use of Powdered (Dry) Infant Formulas in Neonatal Intensive Care Units. Bethesda, MD: US Food and Drug Administration, Center for Food Safety and Applied Nutrition, Office of Nutritional Products, Labeling and Dietary Supplements; 2002.
- [Background] Thoene M, Lyden E, Weishaar K, Elliott E, Wu R, White K, Timm H, Anderson-Berry A. Comparison of a Powdered, Acidified Liquid, and Non-Acidified Liquid Human Milk Fortifier on Clinical Outcomes in Premature Infants. Nutrients. 2016 Jul 26;8(8):451. doi: 10.3390/nu8080451. PMID 27472359
- [Background] Valentine CJ, Morrow G, Reisinger A, Dingess KA, Morrow AL, Rogers LK. Lactational Stage of Pasteurized Human Donor Milk Contributes to Nutrient Limitations for Infants. Nutrients. 2017 Mar 18;9(3):302. doi: 10.3390/nu9030302. PMID 28335478
- See also: Medolac Laboratories — http://www.medolac.com